CLINICAL TRIAL: NCT00921726
Title: Phase 1, Open-Label Study to Evaluate Potential Pharmacokinetic Interactions Between Orally-Administered Oseltamivir and Intravenous Zanamivir in Healthy Thai Adult Subjects
Brief Title: Pharmacokinetic Study of Oseltamivir and Intravenous Zanamivir in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sasithon Pukrittayakamee, MD, Mathidol University, Thailand
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SEA 003
Record Dates: First submitted 2009-06-12; First posted 2009-06-16 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2009-05

CONDITIONS: Influenza; Virus Diseases
Keywords: Drug Interaction
MeSH Terms: conditions — Influenza, Human; Virus Diseases | interventions — Zanamivir; Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive treatment in the following order: Study Regimens A, B, C, D
  Interventions: Drug: Zanamivir; Drug: Oseltamivir
- 2 (Experimental): Participants will receive treatment in the following order: Study Regimens B, A, C, D
  Interventions: Drug: Zanamivir; Drug: Oseltamivir

INTERVENTIONS:
Drug: Zanamivir — Continuous (800 mg in Regimen A, 3600 mg in Regimen C) and intermittent (3600 mg in Regimen D) infusion
  Other Names: Relenza
Drug: Oseltamivir — 150 mg oral tablets taken five times over 3 days in Regimens A, B, C, and D
  Other Names: Tamiflu

SUMMARY:
Due in part to widespread availability of oseltamivir and clinical experience using oseltamivir to treat H5N1 influenza virus infections, many strains of influenza have become resistant to it. Other reliable methods of treating H5N1 must be identified in case of a pandemic. One such option is intravenous zanamivir used in combination with oseltamivir. The primary purpose of this study is to evaluate the interaction between oral oseltamivir and intravenous zanamivir administered as either a continuous or intermittent infusion in healthy adults.

DETAILED DESCRIPTION:
It is very likely that during an influenza pandemic, intravenous zanamivir will be used in combination with oseltamivir. Although the potential for a drug interaction between the two drugs is very low, the likelihood of coadministration combined with the common route of renal clearance of both drugs and the current lack of information on the organic anion transporter polypeptides (OATP) inhibition potential of zanamivir in vivo warrants verification of a lack of an interaction. This study will provide clinical guidance for the use of intravenous zanamivir in settings where oral oseltamivir is commonly used, such as areas in which human cases of H5N1 have been reported.

The total duration of study participation is approximately 13 weeks. Each participant will have a screening visit, four treatment steps, and a follow-up visit. The screening visit to determine enrollment eligibility will be conducted within 45 days prior to receiving the first dose. Participants will be randomized to receive either Regimen A or B for Step 1. Participants who received Regimen A will receive Regimen B in Step 2 and vice versa. After completing Step 2, all participants will continue with Regimens C and D, consecutively, in Steps 3 and 4, with at least 3 days between each step. A follow-up visit will occur 7-10 days after completing the last treatment assessments or withdrawing from the study.

Regimen A consists of continuous intravenous zanamivir infusion (800 mg) for 16 hours. Regimen B consists of 150 mg oral oseltamivir tablets taken five times over 3 days. Regimen C consists of 150 mg oral oseltamivir tablets taken five times over 3 days plus continuous intravenous zanamivir infusion (3600 mg) for 36 hours. Regimen D consists of 150 mg oral oseltamivir tablets taken five times over 3 days plus intermittent intravenous zanamivir infusion received in five 30 minute intervals (3000 mg total).

Blood and urine collection, vital signs, pharmacokinetic sampling, adverse event assessment, and pregnancy test for females will occur at each step in the study. The follow-up visit will involve blood and urine collection, vital signs, adverse event assessment, and pregnancy test for females.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Body mass index between 17 - 32 kg/m^2
* Body weight of at least 37 kg
* Able to read, comprehend, and write at a sufficient level to complete study-related materials
* Normal ECG with QTC less than 450 msec as judged by cardiologist
* Willing and ability to comply with the study protocol for the duration of the trial

Exclusion Criteria:

* History of cardiac disease or abnormality. More information on this criterion can be found in the protocol.
* Family history of sudden cardiac death
* HIV-infected
* Hepatitis C virus infected
* Positive for hepatitis B surface antigen (HBsAg)
* History of renal disease, hepatic disease, and/or cholecystectomy
* Evidence of active substance abuse
* History of alcohol or substance abuse or dependence within 6 months prior to study entry. More information on this criterion can be found in the protocol.
* Use of prescription or non-prescription drugs, except paracetamol, at doses of up to 2 g/day. More information on this criterion can be found in the protocol.
* Use of FluMist, inactivated influenza vaccine, or any other anti-influenza antiviral medications within 14 days prior to study entry
* Participated in a clinical trial and received a drug or new chemical entity within 30 days or five half-lives prior to study entry.
* Unwilling to abstain from ingesting alcohol within 48 hours prior to study entry until collection of the final pharmacokinetic sample during each period
* Donated blood to the extent that participation in this study would result in excess of 300 mL donated within a 30 day period
* History of allergy to the study drug or drugs of this class. More information on this criterion can be found in the protocol.
* Unstable medical condition that, in the opinion of the investigator, would interfere with the study
* Anyone that, in the opinion of the investigator, has a risk of non-compliance with study procedures
* AST or ALN of at least 1.5 ULN
* Certain abnormal laboratory values
* Agree to use effective methods of birth control. More information on this criterion can be found in the protocol.
* Pregnant or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Oseltamivir carboxylate Cmax and AUC (0-12) | Throughout study

SECONDARY OUTCOMES:
Zanamivir Cmax and AUC (0-12) for continuous infusion and Zanamivir Cmax, AUC (-12), and C12 for intermittent infusions | Throughout study
Oseltamivir Cmax, AUC (0-12), and C12 | Throughout study
Oseltamivir carboxylate AUC (0-24), C12, delta-z, and t(1/2) | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Sasithon Pukrittayakamee, MD, Principal Investigator — Mathidol University, Thailand
Locations (1):
- Mathidol University, Salaya, Thailand

REFERENCES:
- [Background] Beigel J, Bray M. Current and future antiviral therapy of severe seasonal and avian influenza. Antiviral Res. 2008 Apr;78(1):91-102. doi: 10.1016/j.antiviral.2008.01.003. Epub 2008 Feb 4. PMID 18328578
- [Background] Hata K, Koseki K, Yamaguchi K, Moriya S, Suzuki Y, Yingsakmongkon S, Hirai G, Sodeoka M, von Itzstein M, Miyagi T. Limited inhibitory effects of oseltamivir and zanamivir on human sialidases. Antimicrob Agents Chemother. 2008 Oct;52(10):3484-91. doi: 10.1128/AAC.00344-08. Epub 2008 Aug 11. PMID 18694948
- [Background] Tappenden P, Jackson R, Cooper K, Rees A, Simpson E, Read R, Nicholson K. Amantadine, oseltamivir and zanamivir for the prophylaxis of influenza (including a review of existing guidance no. 67): a systematic review and economic evaluation. Health Technol Assess. 2009 Feb;13(11):iii, ix-xii, 1-246. doi: 10.3310/hta13110. PMID 19215705